CLINICAL TRIAL: NCT01879267
Title: Exercise Effects in Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2009-0119
Record Dates: First submitted 2012-05-24; First posted 2013-06-17 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training: HD subjects (Other): Endurance exercise for 6 months (30 min per week) starting one week after a 6-months natural course observation
  Interventions: Behavioral: Exercise training
- Exercise Training: healthy subjects (Other): 6 months of exercise training (2 times 30 min per week)
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — 6 months of exercise training (2 times 30 min per week) starting one week after a 6-months natural course observation period

SUMMARY:
Huntington's disease (HD) is an incurable and fatal disorder characterised by progressive degeneration of the basal ganglia and the cerebral cortex. Contrary to earlier thinking, HD is associated with abnormalities in peripheral tissues which might even contribute to brain pathology including muscle wasting, mitochondrial abnormalities, and impaired muscle energy metabolism. Mitochondrial impairment and muscle atrophy in human HD patients and murine models of HD are associated with altered expression of PGC-1a, a transcriptional cofactor that seems to regulate many, if not all of the adaptations of muscle fibres to chronic endurance training, and induces improved exercise performance and increased peak oxygen uptake. We aim at investigating whether endurance exercise has the capability of stabilizing and / or reversing PGC-1a dependent alterations of muscle function and structure in HD patients, and whether muscle training ameliorates musculoskeletal and cardiovascular function, as well as motor and cognitive symptoms in HD patients.

DETAILED DESCRIPTION:
Huntington disease (HD) is an incurable and fatal disorder that affects muscle function and leads to cognitive decline and dementia. HD was long considered a brain disorder but meanwhile it was shown that HD also affects other tissues such as muscle, leading to muscle wasting. Previous studies suggested that the muscle disorder might be caused by an impaired energy metabolism through mitochondrial dysfunction, which also might also contribute to brain pathology.

In muscle tissue of healthy persons, a protein named PGC 1- α seems to regulate many, if not all of the adaptations of muscle metabolism and mitochondrial biogenesis to chronic endurance training. It was shown that PGC 1- α is reduced in muscle tissue of human HD patients and animal models of HD.

We aim investigating whether endurance exercise has the capability of stabilizing and / or reversing PGC-1α dependent decline of muscle function and structure in HD patients, and whether muscle training ameliorates muscular and cardiovascular function, as well as coordination and cognitive decline in HD. To this end, we will train 20 male HD patients using a 6 months progressive endurance exercise program. In order to compare the size effect of exercise between HD patients and healthy individuals, 20 age-matched healthy males will perform the identical exercise regimen as HD patients. Within one week before the training period starts and within one week after it has ended, we will assess metabolic and functional data. In addition, we will analyze muscle tissue samples for muscle fiber structure, metabolic phenotype and cellular pathology. Finally, gene and protein expression analyses will be performed on muscle tissue extracts to gain insights into the molecular regulation of training adaptations in HD.

ELIGIBILITY:
Inclusion criteria: Inclusion criteria for HD subjects are:

* Male gender
* Genetically verified diagnosis of HD
* Age 30 to 50 years
* Presence of only mild to moderate neurological, cognitive or muscular impairment allowing the subjects to give their written informed consent and to participate in the endurance training (UHDRS 30 or lower)

For healthy control participants, inclusion criteria are:

* male gender 9
* age 30 to 50 years
* absence of physical or mental illness

Exclusion criteria: Exclusion criteria for HD subjects are:

* Female gender
* Advanced neurological, cognitive or muscular impairment related to HD that does not allow patients to participate in the endurance training and/or to give their written informed consent
* Cardiovascular disease or any other medical condition that might not be compatible with endurance training
* CK levels > 300 U/L

Exclusion criteria for healthy control participants are:

* cardiovascular disease
* any other medical condition that might not be compatible with endurance training
* CK levels > 300 U/L.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Unified Huntington's Disease Rating Scale (UHDRS) | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Jung, Professor MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Mueller SM, Gehrig SM, Petersen JA, Frese S, Mihaylova V, Ligon-Auer M, Khmara N, Nuoffer JM, Schaller A, Lundby C, Toigo M, Jung HH. Effects of endurance training on skeletal muscle mitochondrial function in Huntington disease patients. Orphanet J Rare Dis. 2017 Dec 19;12(1):184. doi: 10.1186/s13023-017-0740-z. PMID 29258585